CLINICAL TRIAL: NCT01301053
Title: Pilot Study of Intensive Care Unit Continuous Glucose Monitoring
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Virginia (Other)
Collaborators: U.S. Army Medical Research and Development Command (U.S. Federal Agency); University of Texas (Other)
Responsible Party: Principal Investigator, Stacey Anderson, Assistant Professor, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15144
Record Dates: First submitted 2011-02-18; First posted 2011-02-23 (Estimated); Last update posted 2013-01-31 (Estimated); Status verified 2013-01

CONDITIONS: Hyperglycemia; Hypoglycemia
Keywords: hyperglycemia and increased mortality in the ICU; hypoglycemia and increased mortality in the ICU; glucose variability and increased mortality in the ICU; Continuous Glucose Monitoring (CGM) and hypoglycemia; hypoglycemia; reducing ICU mortality
MeSH Terms: conditions — Hyperglycemia; Hypoglycemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Current UVA intensive care insulin protocol without brakes (Other): Studies the safety and feasibility of the continuous glucose monitor in 10 critically ill patients for 7 days and uses the current UVA intensive care insulin for insulin management for 12 hours.
  Interventions: Other: Current UVA intensive care insulin protocol
- Current UVA intensive care insulin protocol with brakes (Active Comparator): Studies the safety and feasibility of the continuous glucose monitor in 10 critically ill patients for 7 days. Uses the current UVA intensive care insulin protocol for insulin management for 12 hours with the addition of "brakes" that reduce insulin administration based on continuous glucose monitoring data between hourly reference glucose data.
  Interventions: Other: Current UVA intensive care insulin protocol with "brakes"

INTERVENTIONS:
Other: Current UVA intensive care insulin protocol — Current UVA intensive care insulin protocol used for insulin management for 12 hours
  Arms: Current UVA intensive care insulin protocol without brakes
Other: Current UVA intensive care insulin protocol with "brakes" — Current UVA intensive care insulin protocol for insulin management with the addition of "brakes" which reduces insulin administration based on continuous glucose monitoring data between hourly reference glucose data to reduce episodes of hypoglycemia (blood glucose <70 mg/dl)and severe hypoglycemia (blood glucose<50 mg/dl).
  Arms: Current UVA intensive care insulin protocol with brakes

SUMMARY:
The investigators believe that there remains a gap in implementing insulin infusions in critically ill patients to maximize the benefit and minimize adverse events like episodes of hypoglycemia. Based on the published experience with Continuous Glucose Monitor (CGM), the investigators believe that it is safe to use in critically ill patients. Furthermore, the investigators believe that in combination with a protocol with low risk for hypoglycemia at baseline, that CGM can eliminate this risk fully.

In this study the investigators will:

1. Study the safety and feasibility of the continuous glucose monitor use in 20 critically ill patients for 7 days (the current maximum recommendation for sensor use). Safety data will include the rate of significant bleeding (hematoma) or infection (cellulitis) from sensor use. Feasibility data will evaluate the amount of missing glucose data over the 7-day sensor life.
2. Randomize patients treated with the current UVA intensive care insulin protocol for insulin management to the addition of "brakes" that reduce insulin administration based on continuous glucose monitoring data between hourly reference glucose data to prevent episodes of hypoglycemia (blood glucose <70 mg/dl) and severe hypoglycemia (blood glucose <50 mg/dl). This will serve as pilot data to power a larger study in the future.

DETAILED DESCRIPTION:
The principle focus of this project is to collect pilot data for a larger study that will test the hypothesis that continuous glucose monitoring (CGM) is safe in critically ill patients and provides important information that can prevent hypoglycemia. This study will determine the feasibility of CGM along with the current UVA intensive care insulin protocol in critically ill hyperglycemic patients as well as to provide some information that may help estimate differences necessary to power future studies.

The following statements summarize the background for this protocol:

1. Hyperglycemia is prevalent in critical illness, even without prior diabetes, and is associated with increased mortality.
2. The physiology between critical illness and hyperglycemia may be secondary to inappropriate tissue oxygenation or intense inflammatory mediator release leading to elevated counter-regulatory hormones that stimulate endogenous glucose production and promote insulin resistance.
3. Early research by Van den Berghe suggested that controlling hyperglycemia by insulin infusion improved outcomes; however, this has been contested in part by the Normoglycemia in Intensive Care Evaluation-Survival Using Glucose Algorithm Regulation (NICE-SUGAR) study.
4. The results of the NICE-SUGAR study may reflect differences in control glucose range or in the high incidence of hypoglycemia.
5. Hypoglycemia has been shown to be associated with increased mortality in the ICU.
6. Glucose variability is associated with ICU mortality.
7. Continuous glucose monitoring has been shown to be safe for up to 7 days in critically ill patients and may prevent episodes of hypoglycemia

ELIGIBILITY:
Inclusion Criteria:

* Age 18 y.o. and above

  * Admitted to an intensive care unit
* Patient will require an insulin infusion or is currently prescribed an insulin infusion during the ICU admission.

Exclusion Criteria:

* Below 18 years of age
* Pregnancy
* Cancer, active diagnosis
* Moribund, Do Not Resuscitate (DNR)/Do Not Intubate (DNI), or death is predicted within 24 hours.
* Patients with diabetic ketoacidosis or hyperosmolar hyperglycemic state will be excluded as they are managed on a different insulin protocol
* Patients with type 1 diabetes will be excluded as they have unique insulin needs that might confound a pilot study.
* Plan for or anticipated need for any MRI during the study period
* Use of acetaminophen within 24 hours prior to enrollment
* Use of a medication on the UVa formulary containing maltose, galactose, or xylose that could affect a glucose dehydrogenase pyrroloquinoline quinine (GDH-PQQ) glucose test strip (hepatitis B immune globulin (HepaGamB®), tositumomab [Bexxar®], abatacept [Orencia®], Octagam 5%, and RH immune globulin [WinRho®])
* Lack of an appropriate abdominal site for insertion of the Dexcom sensor (e.g. extensive scarring, lack of adequate subcutaneous tissue, local infection, etc.)

Restrictions on use of other drugs or treatments.

* According to the Dexcom SEVEN® PLUS and G4 Platinum users manuals, the Dexcom System must be removed prior to Magnetic Resonance Imaging (MRI). Therefore, if the subject requires an MRI, the sensor will be removed from the patient and the reason for removal will be noted. This will not be an Adverse Event, but will conclude the patient's participation in the study.
* If the subject requires the use of acetaminophen-containing medications as part of their clinical care while using the system sensor the subject will be out of the study because this drug may affect the performance of the device.
* If the subject requires use of a medication on the UVa formulary containing maltose, galactose, or xylose that could affect a glucose dehydrogenase pyrroloquinoline quinine (GDH-PQQ) glucose test strip (hepatitis B immune globulin [HepaGamB®], tositumomab [Bexxar®], abatacept [Orencia®], Octagam 5%, and RH immune globulin [WinRho®]) the subject will be out of the study because this drug may affect the performance of the unit glucometer used for reference values and calibration of the continuous glucose monitor. Study participation would be stopped at that time.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2011-02; Primary Completion 2013-09 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
Safety and feasibility of the Continuous Glucose Monitor in critically ill hyperglycemic patients for up to 7 days. | Up to 7 days
  To show that Continuous Glucose Monitor sensors are safe in critically ill patients with a low (<1%) rate of adverse events.

SECONDARY OUTCOMES:
The utility of Continuous Glucose Monitor-driven "brakes" to prevent episodes of hypoglycemia using the current UVA intensive care insulin Protocol | 12 hours
  Continuous Glucose Monitor can prevent episodes of hypoglycemia (defined as a blood glucose less than 70mg/dl) and severe hypoglycemia (defined as a blood glucose less than 50 mg/dl)

CONTACTS AND LOCATIONS:
Overall Officials: Stacey Anderson, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Center for Diabetes Technology, Charlottesville, Virginia, United States